CLINICAL TRIAL: NCT03349749
Title: Does the Use of LiDCOplus Alter Decision-making in Fluid Prescription During Resuscitation in the Intensive Care Unit.
Brief Title: The Use of LiDCOplus in Fluid Resuscitation Decision-Making
Status: Completed | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Other Study IDs: GN16CC090
Record Dates: First submitted 2017-10-25; First posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Shock
Keywords: intensive care units; resuscitation; fluid therapy; Vascular Access Devices; cardiac output; monitoring, physiologic
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing fluid resuscitation: Adult patients in the intensive care unit (ICU) undergoing fluid resuscitation guided by the LiDCOplus haemodynamic monitor.
  Interventions: Device: LiDCOplus haemodynamic monitor

INTERVENTIONS:
Device: LiDCOplus haemodynamic monitor — Patients in study group receive intravenous fluid bolus as part of standard fluid resuscitation. Fluid responsiveness (i.e. improvement in cardiac output) is estimated using both standard clinical parameters and by LiDCOplus haemodynamic monitor (with the clinician initially blinded to the latter) before a final decision about fluid responsiveness is made.

SUMMARY:
Unwell patients in the intensive care unit (ICU) often need supplementary fluids to be given into the bloodstream through a drip in a vein (venous cannula), however too much fluid can be harmful. It can sometimes be difficult to tell whether or not a patient will benefit from extra fluids so they are given a "fluid challenge", whereby a small volume of fluid is given quickly into the cannula and the change in their status is noted. If the patient's condition improves, this suggests that the patient is "fluid responsive" and needs more fluid.

A LiDCOplus haemodynamic monitor is a device used in the ICU to estimate the amount of blood ejected from the heart on each heartbeat using pressure readings obtained from a tube placed in one of the patient's arteries (arterial line).

The investigators aim to determine whether or not the use of this device called makes a difference to the judgement of "fluid responsiveness" when the patient is given a fluid challenge when compared to simply using measurements of pulse and blood pressure and assessing the circulation in the patient's limbs. This will allow the investigators to determine whether or not the LiDCOplus alters the decisions made by doctors and nurses about how much fluid to give their patients and hence if it is of any benefit.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Admitted to Intensive Care Unit (ICU)
* Undergoing fluid resuscitation guided by fluid challenges
* Monitored by a LiDCOplus haemodynamic monitor attached to an arterial line

Exclusion Criteria:

* Poor arterial line trace
* Moribund state
* Patient / relative refusal
* Contra-indication to fluid bolus

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients in the Intensive Care Unit (ICU) undergoing fluid resuscitation guided by fluid challenges monitored by a LiDCOplus haemodynamic monitor.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Fluid responsiveness decisions changed by use of LiDCOplus | 10 minutes
  Proportion of decisions about fluid management changed by knowledge of the change in stroke volume post fluid challenge, as derived by LiDCOplus haemodynamic monitor.

CONTACTS AND LOCATIONS:
Overall Officials: James A Patterson, MBChB, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- Glasgow Royal Infirmary, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/49/NCT03349749/Prot_000.pdf